CLINICAL TRIAL: NCT02578823
Title: Targeted Temperature Management at 36℃ After In-Hospital Cardiac Arrest Trial(TTM36-IHCA Trial): An Investigator-Initiated, Single-Center, Randomized, Controlled, Assessor-Blinded, Pilot Clinical Trial
Brief Title: Targeted Temperature Management After In-Hospital Cardiac Arrest
Acronym: TTM36-IHCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang-Beom Jeon, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-1071
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Targeted Temperature Management(TTM); in-hospital cardiac arrest(IHCA); restoration of spontaneous circulation(ROSC); unconsciousness; brain injury
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Unconsciousness; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TTM-36 (Experimental): Participants assigned to TTM-36 Arm will be managed by Arcticgel™ and Arctic Sun® to maintain core temperatureTemperature at 36.0℃ for 72 hours.
  After targeted temperature management(TTM), Fever will be controlled for remaining 7 days by conventional antipyretic treatment. (Treat core temperature ≥ 38.3℃).
  A total of 40 participants will be enrolled.
  Interventions: Device: Arctic Sun®; Device: Arcticgel™; Procedure: Conventional antipyretic treatment
- Conventional treatment (Active Comparator): Participants who are assigned to this Arm will be treated with conventional antipyretic treatment regarding the occurrence fever for 7 days.(Treat core temperature ≥ 38.3℃).
  A total of 20 participants will be enrolled.
  Interventions: Procedure: Conventional antipyretic treatment

INTERVENTIONS:
Device: Arctic Sun® — Core temperature is maintained to 36℃ for 3 days by using the skin attached pad(Arcticgel™) and targeted temperature management(Arctic Sun®).
  Other Names: Temperature Management System Model 5000
  Arms: TTM-36
Device: Arcticgel™
  Other Names: Hydrogel Coated Pad
  Arms: TTM-36
Procedure: Conventional antipyretic treatment — Conventional antipyretic treatment for fever includes using of antipyretics, ice packs, circulating fan, and tepid bathing, etc.

SUMMARY:
The purpose of this study is to determine whether targeted temperature management at 36.0˚C(TTM-36) in patients who remain unconscious after resuscitation from in-hospital cardiac arrest(IHCA) will reduce death and disability compared with fever control. For this purpose, the current pilot study will be undertaken to establish the feasibility, safety, and surrogate outcomes of hypoxic-ischemic brain injury in 60 patients who remain unconscious after resuscitation from IHCA.

Eligible patients will be randomly assigned in a 2:1 ratio to either TTM-36(n=40) or conventional treatment group(n=20). Randomization will be performed with stratification according to initial rhythm (shockable vs. non-shockable).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* In-hospital cardiac arrest requiring chest compression for > 2 minutes
* Sustained restoration of spontaneous circulation(ROSC) for > 20 minutes after cardiopulmonary resuscitation(CPR)
* Unresponsive state(lack of meaningful response to verbal commands) for > 20 minutes after sustained ROSC
* Informed consents from a patient's family member

Exclusion Criteria:

* Unavailable TTM within 2 hours after ROSC
* CPR duration > 30 minutes
* Unwitnessed arrest with initial rhythm asystole
* Under or planned for extracorporeal membrane oxygenation(ECMO)
* Initial body temperature < 33 °C
* Preexisting terminal illness with life expectancy <6 months
* Pre-admission CPC score of 3-5
* Pre-admission mRS score 4-6
* Unresponsive(stupor or coma) before cardiac arrest
* Suspected or confirmed cause of cardiac arrest is diseases of the central nervous system, such as stroke, brain tumor, or amyotrophic lateral sclerosis
* Any condition in which direct skin surface cooling would be contraindicated, such as large burns, unhealed surgical wounds, decubitus ulcers, cellulitis, or other conditions with disrupted skin integrity
* Active massive bleeding
* Major surgery within last 48 hours
* Cardiothoracic surgery within 14 days
* Planned surgery within next 72 hours after ROSC
* Enrolled in other clinical trials
* Pregnant women
* Do-not-resuscitate(DNR) state
* Patients whose family or treating physicians refuse to join this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Combination of death and poor neurological function defined as a Cerebral Performance Category (CPC) score 3 to 5 at 180 days | day 180
  Efficacy of targeted temperature management at 36.0℃(TTM-36) will be assessed by using Cerebral Performance Category(CPC) score. CPC score is the surrogate outcome for hypoxic-ischemic brain injury.

SECONDARY OUTCOMES:
The CPC score 3 to 5 at day 7 and at day 30 | day 7, day 30
The highest levels of serum neuron specific enolase(NSE) during the first 5 days | up to day 5
Unfavorable Electroencephalography(EEG) patterns | day 0, day 4
  * Generalized suppression(≤20 μV)
  * Burst-suppression with generalized epileptiform activity
  * Generalized periodic epileptiform discharges on a flat background
  * No EEG reactivity
  * Electrographical seizures
  * Electrographical status epilepticus
Assessment of magnetic resonance imaging(MRI) at day 4 | day 4
  * Total magnetic resonance imaging(MRI) scores
  * The percentage of brain volume with Afferent Diffusion Coefficient(ADC) values < 650 x 10^-6mm^2/sec
  * The percentage of brain volume with ADC values < 450 x 10^-6mm^2/sec
  * Number of cerebral microbleeds
Modified Rankin Scale(mRS) score 4 to 6 at day 30 and at Day 180 | day 30, day 180
All-cause mortality at day 30, at Day 180 | up to day 180
Myoclonic or tonic-clonic seizures or status epilepticus(SE) | up to day 7
Neurological status estimated by the Seoul Neurosychological Screeninig Battery (SNSB) 2nd ed. | day 180
  * Attention: Digit span (forward), digit span (backward)
  * Language & related function: Spontaneous speech, comprehension, repetition, reading, writing, finger naming, body part identification, right-left orientation, calculation; BNT (Boston Naming Test)
  * Visuospatial: RCFT (Rey Complex Figure Test) copy score
  * Memory: SVLT (Seoul Verbal Learning Test), RCFT (immediate recall, delayed recall, recognition)
  * Frontal & executive function: COWAT (Controlled Oral Word Association Test), CWST (Color Word Stroop Test), DSC (Digit Symbol Coding), TMT (Trail making test)
  * General cognitive index: MMSE (Mini Mental State Examination), CDR (Clinical Dementia Rating), GDS (Global Deterioration Scale)
  * Activities of daily living (ADL): Barthel index
Other neurological evaluations | day 180
  * Depression: BDI (Beck Depression Inventory)
  * Quality of life: SF-36 (Short-Form 36-item Health Survey)
  * Activities of daily life: S-IADL (Seoul-Instrumental Activities of Daily Living)
  * Psychiatric symptoms: NPI (Neuropsychiatric Inventory)
  * Cognition: IQCODE (Informant Questionnaire on Cognitive Decline in the Elderly)
  * Parkinsonism: UPDRS (Unified Parkinson's Disease Rating Scale)
  * Ataxia: ICARS (International Cooperative Ataxia Rating Scale)
Assessment of follow-up MRI | day 30 & day 180
  * Resting state functional MRI: Connectivity strength, proportional increase of connectivity strength on resting state
  * Diffusion tensor imaging: Global mean diffusivity, gray matter mean diffusivity, white matter mean diffusivity , mean fractional anisotropy, proportional increase of white matter global fractional anisotropy, proportional increase of white matter global mean diffusivity
  * High resolution T1-weighted imaging for MRI volumetric: Mean volume of the brain, mean volume of the gray matter of the brain, mean volume of the white matter of the brain, proportional increase of mean volume of the brain, proportional increase of mean volume of the gray matter, proportional increase of mean volume of the white matter
  * Susceptibility-weighted imaging: Number of cerebral microbleeds

OTHER OUTCOMES:
Safety of the targeted temperature management at 36.0℃(TTM-36) | up to day 7
  Safety will be assessed by the composite measurement below everyday during the first 7 days after cardiac arrest.
  * Cardiac arrest after randomization
  * Arrhythmia(ventricular fibrillation, ventricular tachycardia, atrial fibrillation, atrial flutter, tachycardia >130/min lasting more than 1 hour, and bradycardia <40/min lasting more than 1 hour)
  * Pneumonia(pulmonary infiltration on the chest radiography and 2 or more of fever, leukocytosis, and purulent tracheobronchial secretions)
  * Septic shock(sepsis-induced hypotension persisting despite adequate fluid resuscitation)
  * Culture-proven infection
  * Major bleeding(bleeding requiring more than 2 units of packed red blood cell over 2 hours, bleeding causing fatality, and symptomatic bleeding in critical organs)
  * Shivering(the Bedside Shivering Assessment Scale 2-3)
Feasibility | up to day 180
  * 2.5 subjects per month can be recruited
  * At least 50% of all eligible patients can be recruited
  * No more than 10% of all recruited subjects cross over from one modality to the other
  * Complete follow-up in at least 90% of all recruited subjects

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Beom Jeon, Dr, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea